CLINICAL TRIAL: NCT02050685
Title: Comparison of Different Screening Score for Hypoxemic OSA
Brief Title: Comparison of Different Screening Score for Hypoxemic OSA (Obstructive Sleep Apnea) With the Results of a Polysomnography (PSG)
Status: Completed | Type: Observational
Sponsor: Eric DEFLANDRE, MD, FCCP (Other)
Responsible Party: Sponsor-Investigator, Eric DEFLANDRE, MD, FCCP, ERIC DEFLANDRE, MD, FCCP, Astes
Organization: Astes (Other)
Other Study IDs: REES-ASTES-2014
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients for PSG at SLBO: All patients incoming in the sleep study centre for a PSG. At the arrival the screening score will be recorder. AHI will be recorded next morning after analysis of the PSG.
  Interventions: Other: All patients incoming in the sleep study centre for a PSG

INTERVENTIONS:
Other: All patients incoming in the sleep study centre for a PSG — All patients incoming in the sleep study centre for a PSG. Comparison between screening score and AHI derived from PSG.

SUMMARY:
Comparison of different screening score for hypoxemic OSA (Obstructive Sleep Apnea) with the results of a polysomnography (PSG). The different screening score studied are: STOP-BANG, DES-OSA, P-SAP and OSA50.

DETAILED DESCRIPTION:
The investigators should compare the four screening scores (STOP-BANG, DES-OSA, P-SAP and OSA50) with the results of the PSG (and in particular the number of apnea and hypopnea index and the probability of hypoxemia).

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (> 18 years)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults patients for an overnight polysomnography at SLBO.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the DES-OSA score with previously described scores. | The day before the PSG (PolySomnoGraphy)
  Comparison of the DES-OSA score with the results of previously described scores (STOP-BANG, P-SAP and OSA50).

SECONDARY OUTCOMES:
Comparison of the four screening scores with results of the PSG. | The day after the polysomnography
  Comparison of the four screening scores collected past day (before PSG - PolySomnoGraphy) with the results of the PSG (especially the AHI: Apnea Hypopnea Index)

CONTACTS AND LOCATIONS:
Overall Officials: Eric P DEFLANDRE, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc de Bouge, Bouge, Namur, Belgium

REFERENCES:
- [Derived] Deflandre E, Piette N, Bonhomme V, Degey S, Cambron L, Poirrier R, Brichant JF, Joris J. Comparison of clinical scores in their ability to detect hypoxemic severe OSA patients. PLoS One. 2018 May 7;13(5):e0196270. doi: 10.1371/journal.pone.0196270. eCollection 2018. PMID 29734398